CLINICAL TRIAL: NCT03998176
Title: A Phase 4, Single-Arm Study of the Efficacy and Safety of Bictegravir/Emtricitabine/Tenofovir Alafenamide in HIV-1 Infected Patients With Active Illicit Substance Use
Brief Title: Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF) in HIV-1 Infected Patients With Active Illicit Substance usE
Acronym: BASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0471-19-FB
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: HIV-1-infection
Keywords: Substance use
MeSH Terms: conditions — Substance-Related Disorders | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- B/F/TAF (Experimental): Participants will receive B/F/TAF for 48 weeks
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide

INTERVENTIONS:
Drug: Bictegravir/emtricitabine/tenofovir alafenamide — B/F/TAF single tablet formulation
  Other Names: Biktarvy

SUMMARY:
This study will evaluate the efficacy and safety of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) in HIV-1 infected patients who actively use illicit substances. The study will also evaluate retention in care and adherence to B/F/TAF by self-report and pharmacokinetic analysis.

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective, pilot study to evaluate the effectiveness and safety of B/F/TAF in viremic HIV-1 infected treatment naive or experienced patients with active illicit substance use outside of nicotine, alcohol, and marijuana use.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Treatment naive or experienced
* Self-reported illicit substance use or confirmed urine drug screen within past 6 months of any of the following: cocaine, heroin, methamphetamine, MDMA, phencyclidine, ketamine, gamma hydroxybutyrate, cathiniones, or inappropriate prescription opiate, benzodiazepine or stimulant use (excluding nicotine, alcohol, marijuana for criteria)
* HIV RNA >1000 copies/mL
* Creatinine clearance > 30 mL/min (Cockroft-Gault)
* ALT and AST < 5 times the upper limit of normal
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of integrase or tenofovir related HIV resistance mutations
* Pregnancy
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Havens, PharmD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B/F/TAF: Daily through week 48
Period: Overall Study
Arm/Group | B/F/TAF
Started | 43
Completed | 31
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: All 43 participants received 1 dose of B/F/TAF and are included in the intent-to-treat analysis.
Arm/Group | B/F/TAF
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [21 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL as Determined by the FDA-defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24 analyzed by the snapshot algorithm, which defines a participants virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 43
Participants | 32

2. Secondary Outcome: Percentage of Participants With Grade 3 or Greater Adverse Events
Description: The percentage of participants experiencing grade 3 or greater adverse events at Week 24
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 43
Participants | 12

3. Secondary Outcome: Percentage of Participants With Grade 3 or Greater Adverse Events
Description: The percentage of participants experiencing grade 3 or greater adverse events at Week 48
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 43
Participants | 15

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL as Determined by the FDA-defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 analyzed by the snapshot algorithm, which defines a participants virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 43
Participants | 21

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | B/F/TAF
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 15/43
Other Adverse Events (participants affected / at risk) | 5/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B/F/TAF (N=43)
Grade 3 or above SAE (Investigations) | 15 (27) — According to DAIDS AE Grading Table
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B/F/TAF (N=43)
Suicidal Ideation (Psychiatric disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03998176/Prot_SAP_000.pdf